CLINICAL TRIAL: NCT01443481
Title: A Multi-center, Open Label Study to Assess Pharmacokinetics of TKI258 in Adult Cancer Patients With Normal and Impaired Hepatic Function
Brief Title: Pharmacokinetics (PK) of TKI258 in Cancer Patients With Normal and Impaired Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTKI258A2124; 2011-000103-41 (EudraCT Number)
Record Dates: First submitted 2011-09-17; First posted 2011-09-29 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2017-06

CONDITIONS: Solid Tumors; Hepatic Impairment
Keywords: solid tumors; hepatic impairment; Child-Pugh classification; pharmacokinetics; PK; RECIST 1.1
MeSH Terms: interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- TKI258 normal hepatic function (Experimental): TKI258 Capsule, @ 500 mg p.o. o.d. 5 days on/2 days off
  Interventions: Drug: Dovitinib
- TKI258 mild hepatic impairment (Experimental): TKI258 capsule @ 500 or 400 mg p.o. o.d. 5 days on/2 days off
  Interventions: Drug: Dovitinib
- TKI258 moderate hepatic impairment (Experimental): TKI258 capsule @ starting dose at 400 mg p.o. o.d. 5 days on/2 days off
  Interventions: Drug: Dovitinib
- TKI258 severe hepatic impairment (Experimental): TKI258 capsule Starting dose to be determined based on the study outcome of the mild and moderate hepatic impairment groups
  Interventions: Drug: Dovitinib

INTERVENTIONS:
Drug: Dovitinib — Starting dose to be determined based on the study outcome of the mild and moderate hepatic impairment groups
  Other Names: TKI258

SUMMARY:
This is a multi-center, open label study to assess pharmacokinetics (PK) of TKI258 at single-dose and steady state in adult cancer patients either with mild, moderate or severe hepatic impairment or with normal hepatic function. Hepatic function in study patients will be categorized as normal, mild, moderate or severe based upon pre-dose (Day 1) total bilirubin and AST/ALT levels. Starting dose of TKI258 will depend on total bilirubin and ALT/AST levels at baseline. Patients will be treated until disease progression (assessed by RECIST 1.1), unacceptable toxicity, death or discontinuation from the study treatment for any other reason.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically or cytologically confirmed solid tumor, excluding breast cancer, that is either refractory to the standard therapy or has no available therapies.
2. ECOG performance status (PS) 0 or 1
3. Patients must have measurable and/or non-measurable lesion(s) as assessed by Computer Tomography (CT) Scan or Magnetic Resonance Imaging (MRI) per RECIST 1.1

Exclusion Criteria:

1. Patients with known brain metastases.
2. Patients who have undergone major surgery ≤ 4 weeks prior to starting study treatment

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2011-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) parameter of Cmax following a single dose of TKI258 and at the steady state | Day 1, Day 19
  Cmax will be evaluated after a single dose of TKI258 and at the steady state following a 5 days on/2 days off dosing schedule. Cmax is the maximum (peak) plasma, blood, serum, or other body fluid drug concentration after a single dose administration (mass x volume - 1).
Pharmacokinetic (PK) parameter of Tmax following a single dose of TKI258 and at the steady state | Day 1, Day 19
  Tmax will be evaluated after a single dose of TKI258 and at the steady state following a 5 days on/2 days off dosing schedule. Tmax is the time to to reach maximum (peak) plasma, blood, serum, or other body fluid drug concentration after a single dose administration (mass x volume - 1).
Pharmacokinetic (PK) parameter of AUClast following a single dose of TKI258 and at steady state | Day 1, Day 19
  AUClast will be evaluated after a single dose of TKI258 and at the steady state following a 5 days on/2 days off dosing schedule. AUC from time zero to the last measurable concentration sampling time t(last) (mass x time x volume^-1)
Pharmacokinetic (PK) parameter of AUCinf following a single dose of TKI258 | Day 1, Day 19
  AUCinf is the time to zero to infinity (mass x time x volume)

SECONDARY OUTCOMES:
Frequency of Adverse Events and Serious Adverse Events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) | Baseline and every 4 weeks
  The Common Terminology Criteria for Adverse Events (AE) is a descriptive terminology which can be utilized for AE reporting. An AE is any unfavorable and unintended sign (including an abnormal laboratory finding),symptom, or disease temporally associated with the use of a treatment.
Change from Baseline in Vital Signs | Baseline, Weeks 1, 4, 5, 9 and once every 8 weeks thereafter
  Body temperature, sitting pulse rate, and sitting blood pressure will be measured at each visit. Blood Pressure (BP) will be measured according to the National Institute of Health, National Hart, Lung and Blood Institute Guidelines with following standardized techniques: patients are seated; BP measurement begins after at least 5 minutes of rest, the appropriate cuff size is used , measurements will be taken preferably with a mercury sphygmomanometer. If the BP reading is ≥ 160mm Hg systolic and/or ≥100 mmHg diastolic, repeat the measurement to verify initial reading.
Best overall response to anti-tumor activity of TKI258 through imaging as per RECIST 1.1 | Every 8 weeks
  RECIST (Response Evaluation Criteria In Solid Tumors) is a set of published rules that define when cancer patients improve ("respond"), stay the same ("stable") or worsen ("progression") during treatments.
Change from Baseline in Electrocardiogram | Baseline, Weeks 1, 4, 5
  A standard 12 lead Electrocardiogram(ECG)will be used. In order for an accurate evaluation of baseline QTc, a total of three 12-lead ECGs will be performed within 72 hours prior to the first dose of TKI258 administration on Week 1, Day 1. All ECGs will be transmitted to a central laboratory and will be centrally reviewed by an independent reviewer.
Pharmacokinetics and Hepatic Function Abnormalities | Baseline, every 4 weeks
  Exploration of the relationship between Pharmacokinetics (PK) and hepatic functional abnormalities (i.e. bilirubin, ALT/AST, and Child-Pugh classification using regression analysis as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- United States (3):
  - University of California at Los Angeles Dept. of UCLA (4), Los Angeles, California
  - Duke University Medical Center DUMC, Durham, North Carolina
  - Cancer Therapy & Research Center / UT Health Science Center SC, San Antonio, Texas
- Novartis Investigative Site, Ghent, Belgium
- Germany (2):
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Hanover
- Italy (3):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Verona, VR
- Netherlands (2):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Maastricht
- Novartis Investigative Site, Singapore, Singapore

REFERENCES:
- See also: Results for CTKI258A2124 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=13906